CLINICAL TRIAL: NCT04978220
Title: Follow-up Study on Mental and Psychological Problems and Insomnia Disorder of Medical Staff in Hospital Where Staff Are Infected With COVID-19
Brief Title: Mental and Psychological Problems and Insomnia Disorder of Medical Staff in Hospital With Infected COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Xueqin Wang, Principle Investigator, Peking University Sixth Hospital
Other Study IDs: 2020-021(BMR)
Record Dates: First submitted 2021-07-19; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Depression Unipolar; Insomnia
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to clarify the severity of psychological problems and insomnia and the two's relationship with time of hospital medical staff in hospital where its staff are infected with COVID-19.

DETAILED DESCRIPTION:
A cross-sectional questionnaire survey method was adopted to conduct investigations of medical staff in the researched hospital within one week (baseline) and one year (follow-up) after the discovery of COVID-19 infection cases. 360 subjects were included in the baseline. Then, after one year, 199 subjects who participated in the survey at baseline were included as follow-up. The HADS, ASDS and ISI scales were used to assess the anxiety and depression level, acute stress disorder symptoms, and the severity of insomnia of hospital medical staff; self-made questionnaires was to collect demographic information and descriptive content. Comparing the follow-up medical staff with the baseline, the total scores of ASDS, HADS and ISI, each item scores on the ASDS, HADS and ISI. All of above scales are compared between the quarantined and non-quarantined groups, different quarantined groups (home, hotel, hospital) and non-quarantined groups.

ELIGIBILITY:
Inclusion Criteria:

* all medical staff of a third-level general hospital in Beijing who discovered a sporadic case of COVID-19 infection; Volunteer to participate in surveys and follow-ups

Exclusion Criteria:

* Incomplete information fills in, which affects the result analysis

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were 644 medical staff on duty in the hospital, of which 360 people participated in the baseline survey, accounting for 55.90%. In the follow-up survey after one year, 199 out of 360 people in the baseline participated, accounting for 55.28% of the baseline.
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 1 year
  HADS is used to assess the anxiety and depression symptoms of medical staff in general hospitals. There are 14 items in total, divided into two parts-the anxiety subscale (HADS-A) and the depression subscale (HADS-D). A total score of 0-7 is classified as asymptomatic, 8-10 is classified as marginal/suspicious, and 11-21 is classified as abnormal.

SECONDARY OUTCOMES:
Acute Stress Disorder Scale (ASDS) | 1 year
  ASDS is a self-rating scale, compiled according to the diagnostic criteria of the fourth edition of the "Manual of Diagnosis and Statistics of Mental Disorders", used to assess acute stress disorder (ASD) symptoms and predict post-traumatic stress disorder (PTSD).

OTHER OUTCOMES:
Insomnia Severity Index (Insomnia Severity Index, ISI) | 1 year
  ISI is a simple tool for screening insomnia, including 7 items to assess the severity of the subjects' sleep symptoms, the subjects' satisfaction with their sleep patterns, the impact of the degree of insomnia on daily functions, the subjects' awareness of the impact of insomnia on themselves, and the level of depression caused by sleep disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqin Wang, MD, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No